CLINICAL TRIAL: NCT03588689
Title: Continuous Fascia Iliaca Block for Acute Hip Fractures: a Randomized Controlled Pilot Study
Brief Title: Continuous Fascia Iliaca Block for Acute Hip Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Churao Yang, Anesthesiologist, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bio 17-267
Record Dates: First submitted 2018-04-27; First posted 2018-07-17 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Hip Fractures; Neuromuscular Blockade; Respiratory Morbidity; Delirium; Fascia Iliaca Block; Pain
Keywords: hip fracture; fascia iliaca block; continuous fascia iliaca block; neuromuscular blockade
MeSH Terms: conditions — Hip Fractures; Delirium; Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: This study is a prospective randomized controlled non-blinded pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Treatment (No Intervention): Patients in this group will receive standard treatment orders which include a combination of opioids, NSAIDs, acetaminophen, and other adjuncts for analgesia.
- Continuous fascia iliaca block (Experimental): The cFIB group will receive an ultrasound guided cFIB and standard treatment orders as backup in the event of block failure.
  The cFIB group will receive an initial bolus of 40 cc of 0.25% Ropivacaine followed by an infusion of 8 cc/hr until the time of surgery. Immediately pre-operatively, the anesthesiologist performing the case will bolus the catheter 40 cc of 0.25% ropivacaine and discontinue the catheter.
  Interventions: Procedure: Continuous fascia iliaca block; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Continuous fascia iliaca block — Regional nerve block performed under ultrasound guidance. A catheter will be left in place to allow ongoing infusion of local anesthetic.
  Arms: Continuous fascia iliaca block
Drug: Ropivacaine — Ropivacaine local anesthetic will be used for the fascia iliaca block
  Arms: Continuous fascia iliaca block

SUMMARY:
Hip fractures are a major cause of morbidity and mortality in the elderly with over 30,000 hip fractures occuring in Canada annually and over 1300 in Saskatchewan. The estimated cost associated with hip fractures is over $600 million nationally and 28 million dollars in Saskatchewan. Hip fractures cause a great deal of pain and immobility and are mainly treated with surgical fixation. In the perioperative period, hip fracture patients are treated mainly with opioids and other adjuncts such as NSAIDS and acetaminophen. Opioid consumption in the elderly population can predispose to delirium and respiratory complications such as atelectasis, respiratory depression, and pneumonia.

Fascia iliaca blocks have been shown to be an effective mode of analgesia for patients with hip fractures, but are underutilized for varying reasons including culture of practice, expertise with performing the block, and having a dedicated service to do so.

This study aims to compare the efficacy of fascia iliaca blocks to standard treatment (opioids) in the management of pain in hip fracture patients with a particular focus on outcomes such as the incidence of delirium, respiratory complications, and length of stay in hospital. Our idea is that if we can reduce the amount of opioids these patients receive then they will have improved pain control, fewer respiratory complications, earlier time to mobilizing, and shorter hospital stays. As far as we are aware this relation has not been well studied.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled non-blinded pilot study.

Recruitment and Randomization: fifty adult patients with hip fractures for surgical fixation presenting to Royal University Hospital (RUH), Saskatoon, Saskatchewan, will be recruited. The exclusion criteria are:

* American Society of Anesthesiologists (ASA) score >3
* Other injuries that interfere with block positioning and assessment of pain
* Local anesthetic allergy
* Open fracture
* Moderate to severe pre-operative delirium (interfering with consent and assessment)
* Sepsis at site of injection
* Anticoagulation with warfarin or anti-Xa inhibitors
* Age less than 65 years

Patients will be randomized into one of two research arms: Continuous Fascia Iliaca block (cFIB) vs standard treatment (opioids). It is important to note here is that patients receiving cFIBs will have standard treatment orders available in the event of block failure, and opioid consumption will be monitored.

Methods:

Patients with hip fractures presenting to RUH will be approached by a member of the study team for consent to participate in the study. After consent is obtained patients will be randomised to either arm of the study group. The cFIB group will receive an ultrasound guided cFIB and standard treatment orders as backup in the event of block failure. The standard treatment group will receive only standard treatment orders which include a combination of opioids, NSAIDS, acetaminophen, and other adjuncts for analgesia.

The CFIB group will receive an initial bolus of 40 cc of 0.125% Ropivacaine followed by an infusion of 10 cc/hr of 0.2% ropivacaine until the time of surgery. Immediately pre-operatively, the anesthesiologist performing the case will bolus the catheter with 40 cc of 0.125% ropivacaine and discontinue the catheter.

Data collection: Demographic and epidemiologic data will be collected for both groups at the time of recruitment. Patients will be followed from the time of enrollment until the time of discharge from hospital. A member of the study team will visit daily and assess the patients for delirium using the Confusion Assessment Method (CAM)-ICU tool, which is a validated delirium assessment tool. Pain scores will be obtained after block insertion and twice a day until surgical fixation takes place. Pain scores will be assessed in the supine, semi recumbent, and upright position, and with active movement. Opioid consumption will be recorded as morphine equivalents for the entire length of hospital stay. The incidence of side effects of opioids will be recorded including : Nausea, vomiting, pruritis, constipation, and urinary retention.

The length of time from surgery until ready to discharge will be recorded.

It is difficult to directly measure respiratory complications. As a surrogate for respiratory complications the following data will be collected:

* Oxygen requirements pre and post operatively
* Pre and post operative need for positive pressure ventilation (CPAP, BiPAP)
* Radiographic evidence of atelectasis or pneumonia
* Trends in oxygen saturation as measured by pulse oximetry Data collection is projected to be completed by July 1st 2018

Data analysis: Parametric data will be reported as a mean +/- standard deviation, along with confidence intervals. Means will be used to estimate effect size and these values will then be used in power calculations and sample size estimation for future studies. In addition, the unpaired t-test will be used to test for significant difference between groups. The incidence of adverse events will be recorded and presented with descriptive statistics. Data analysis is projected to be completed by October 2018

Significance:

Fascia Iliaca blocks have already been shown to improve pain in hip fracture patents. Our theory is that if we can effectively manage pain with cFIBs we can reduce the amount of opioids patients receive in the perioperative period. This could lead to reduced complications from opioids, improved patient positioning, improved patient mobility, and earlier time to discharge which would have a great impact on patient experience and cost of care.

ELIGIBILITY:
Inclusion Criteria:

* Adults age greater than or equal to 65 years old with acute hip fracture

Exclusion Criteria:

* ASA greater than or equal to 4
* Open fractures
* Other concomitant injuries that may interfere with positioning or pain scores
* Local anesthetic allergy
* Delirium at the time of consent
* Pre-existing cognitive impairment
* Infection at the site of injection for cFIB
* Previous surgery in femoral triangle
* Warfarin or Anti-Xa inhibitor use
* Long-term opioid use
* Intraoperative complications

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Respiratory complications | During hospital stay, up to 1 month
  Use of supplemental oxygen, need for positive pressure ventilation, decreased oxygen saturations, radiographic evidence of atelectasis or pneumonia

SECONDARY OUTCOMES:
Pain score | During hospital stay, up to 1 month
  Subjective pain score on 1-10 visual analog scale in supine, semi-recumbent, upright positions, and with active movement
Opioid side effects | During hospital stay, up to 1 month
  Incidence of nausea, vomiting, pruritus, constipation, and urinary retention will be recorded
30 day mortality | Will be collected from hospital record, at up to 3 months after enrolment.
  Status, living or deceased, at 30 days post op
Delirium | During hospital stay, up to 1 month
  CAM-ICU scoring system will be used daily to measure delirium
Post op length of stay | During hospital stay, up to 1 month
  Will be measured as number of days in hospital from date of admission until ready for discharge

CONTACTS AND LOCATIONS:
Overall Officials: Brian Brownbridge, MD, Principal Investigator — University of Saskatchewan; Churao Yang, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data.

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043